CLINICAL TRIAL: NCT03759353
Title: A Comparative Study Between Lactoferrin Versus Ferrous Sulfate in Iron-deficiency During Pregnancy
Brief Title: Lactoferrin Versus Ferrous Sulfate in Iron-deficiency During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Ahmed, Resident of O&G, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LactvsFerr
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; ferrous sulfate; Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: 98 pregnant women with iron deficiency will be randomized into two groups: lactoferrin group or ferrous sulfate group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin Group (Active Comparator): Includes 49 pregnant women receiving lactoferrin 100 mg one sachet twice daily for 30 days to be dissolved in 1/4 glass of water before meals (Pravotin (R) , Hygint pharmaceuticals). Baseline ferritin level will be obtained and compared to follow up ferritin level after 30 days of treatment.
  Interventions: Diagnostic Test: Baseline ferritin level; Drug: Lactoferrin; Diagnostic Test: Follow up ferritin level
- Ferrous Sulfate Group (Active Comparator): Includes 49 pregnant women receiving 200 mg of dried ferrous sulfate tablet once daily for 30 days on empty stomach but may be taken with meals to avoid stomach upset (Feosol (R) , Meda pharmaceuticals). Baseline ferritin level will be obtained and compared to follow up ferritin level after 30 days of treatment.
  Interventions: Diagnostic Test: Baseline ferritin level; Drug: Ferrous Sulfate; Diagnostic Test: Follow up ferritin level

INTERVENTIONS:
Diagnostic Test: Baseline ferritin level — At enrollment, baseline serum ferritin level will be assessed to quantify iron deficiency.
Drug: Lactoferrin — lactoferrin 100 mg one sachet twice daily for 30 days to be dissolved in 1/4 glass of water before meals (Pravotin, Hygint pharmaceuticals).
  Other Names: Pravotin
  Arms: Lactoferrin Group
Drug: Ferrous Sulfate — 200 mg of dried ferrous sulphate tablet once daily for 30 days on empty stomach but may be taken with meals to avoid stomach upset.
  Other Names: Feosol
  Arms: Ferrous Sulfate Group
Diagnostic Test: Follow up ferritin level — Four weeks after treatment, serum ferritin level will be assessed to quantify effect if treatment on iron status.

SUMMARY:
The main drawbacks with oral iron are side-effects, poor compliance, and limited absorption from the gut. It has become very apparent gastrointestinal intolerance with oral iron therapy is dose related and common (up to 20% of patients), and this frequently leads to poor compliance.

Lactoferrin (formerly known as lactotransferrin) is a glycoprotein, and a member of a transferrin family, thus belonging to those proteins capable of binding and transferring iron. It represents an attractive and promising alternative to ferrous sulphate oral administration as pregnant women receiving lactoferrin did not experience any adverse effects.

This study aims to compare between lactoferrin and ferrous sulphate for therapy of iron deficiency in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with single fetus.
* Second trimester (14-20weeks of gestation).
* Normal Hemoglobin level: more than10g\dl.
* Serum ferritin less than 15 mcg / L

Exclusion Criteria:

* Other type than iron-deficiency anemia (thalassemia, hemolytic anemia … etc.)
* Any other chronic diseases (bronchial asthma, renal or hepatic, hematological or cardiovascular diseases … etc.)
* Having hypersensitivity to iron preparations.
* Treatment with any other iron preparation in the last month.
* History of peptic ulcer, oesophagitis or hiatal hernia.
* Medical disorders with pregnancy.
* Need for alternative parenteral route to blood transfusion when rapid increase is required (perioperative anemia-severe anemia in late pregnancy-postpartum anemia) .
* Bleeding in early pregnancy.
* Refusal to participate in the study.
* Family history of thalassemia-sickle cell anemia or malabsorption syndrome.
* Recent blood transfusion.
* Inflammatory bowel disease as intolerance of oral therapy but tolerated to parenteral route.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin level | 4 weeks
  Change in serum ferritin level between enrollment and 4 weeks post-treatment.

SECONDARY OUTCOMES:
Nausea and/or vomiting | 4 weeks
  Incidence of treatment-related nausea and/or vomiting
Dyspepsia | 4 weeks
  Incidence of treatment-related dyspepsia
Compliance to treatment | 4 weeks
  Number of missed doses of treatment from the assigned 30 doses

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Mohamed, MBBCh, Principal Investigator — G Darwish
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No